CLINICAL TRIAL: NCT01994174
Title: Effect of Vascular Endothelial Growth Factor Blockers on Aqueous Humor Dynamics
Status: Terminated | Type: Observational
Why Stopped: Limited resources; IRB approval was not maintained
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0583-13-FB
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Macular Disease
Keywords: vascular; retina; Anti-VEGF; Aqueous humor dynamics
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this research is to determine the effects of anti-VEGF drugs (bevacizumab, ranibizumab or aflibercept) on aqueous humor dynamics (AHD) in patients with retinal vascular disease. The underlying hypothesis is that anti-VEGF drugs increase intraocular pressure (IOP) by increasing aqueous inflow, decreasing uveoscleral outflow or both. The specific aim is to evaluate the changes produced in AHD after 1 baseline and a subsequent 1 monthly injection of anti VEGF agents.

DETAILED DESCRIPTION:
Intravitreal injection of different anti-VEGF agents such as bevacizumab (Avastin, Genentech, Inc., South San Francisco, CA, USA) ranibizumab (Lucentis; Genentech, Inc., South San Francisco, CA, USA) and aflibercept (Eylea, Regeneron, Tarrytown, NY, USA) has been a widely common practice for treatment of choroidal neovascularization and retinal vascular diseases [1]. Several ocular and systemic adverse events have been reported with the use of anti-VEGF agents [7]. Elevation of intraocular pressure (IOP) is a serious ocular adverse event that may be associated with intravitreal injection of anti-VEGF agents. IOP elevation with anti-VEGF injection may have variable presentation ranging from acute transient post injection elevation to the development of persistent IOP elevation that mandates pressure lowering therapy[8].

Patients with previously existing glaucoma may have a higher rate of persistent IOP elevation associated with intravitreal injection of anti-VEGF agents. Good et al, reported the rate of persistent IOP elevation after intravitreal anti-VEGF to be 33% in glaucoma patients versus 3.1% in eyes without previous diagnosis of glaucoma [9]. Tseng et al, reported 25 eyes with sustained elevation of IOP after serial intravitreal injections of anti-VEGF agents (mean = 20injections). All the 25 eyes were normotensive prior to the study and 23 of them were not previously diagnosed with glaucoma[10].

Multicenter clinical trials that studied the intravitreal injection of anti-VEGF agents, such as MARINA and ANCHOR for ranibizumab, VISION for pegaptanib and PACORES for bevacizumab, did not show sustained IOP elevation with the intravitreal injection of the study agents [12-15]. However, a subgroup analysis of the data of MARINA and ANCHOR trials showed at least 6 mm Hg increase of IOP from baseline in 2.1% of eyes in MARINA trial and 3.6% of eyes in ANCHOR trial [16]. A retrospective chart review of 207 patients over a 6-months follow up period after serial intravitreal injections of anti-VEGF reported an IOP elevation greater than 5 mm Hg in 2 consecutive visits compared to baseline in 11.6% of the treated eyes versus 5.3% in control eyes [17].

The pathophysiology of the reported IOP elevation associated with intravitreal injection of anti-VEGF is unknown. Anti-VEGF compounds might increase aqueous humor inflow by the breakdown of the blood-aqueous barrier or reduce uveoscleral outflow by the ciliary body vasculature. These potential changes could translate into elevated IOP and glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 19 years of age and older
* Ability to give informed consent and attend the study visits
* Patients with established diagnosis of retinal vascular diseases (diabetic macular edema, neovascular macular degeneration,presumed ocular histoplasmosis syndrome, high myopia) who require intravitreal injection of anti-VEGF drugs such as bevacizumab,ranibizumab or aflibercept and are likely to need three monthly doses.
* Patients who have not received intravitreal injections within 3 months of study entry
* No previous established diagnosis of glaucoma and consequently no previous history of Argon Laser Trabeculoplasty (ALT) or Selective Laser Trabeculoplasty (SLT).
* No previous history of ocular surgery
* Patients who are not planning on and are unlikely to require an elective ocular surgical or laser procedure within the study duration
* Open angle of the anterior chamber on clinical examination
* Ability to cooperate for aqueous humor dynamic studies
* Contact lenses removed prior to topical fluorescein instillation, and not used until the end of each fluorophotometry session
* Able to participate on site over the multi-visit study period

Exclusion Criteria:

* Age less than 18 years of age
* Women who are pregnant or nursing
* Ocular hypertension or glaucoma
* Narrow angle with complete or partial closure (gonioscopy angle <2)
* Any previous surgical or laser procedures
* Secondary glaucoma including pigmentary, exfoliative, uveitic and traumatic glaucomas
* Any active neovascularization of the iris, angle, disc or retina
* Diagnosis of retinal arterial or vein occlusion
* Chronic or recurrent inflammatory eye disease
* Ocular trauma within the past 6 months
* Ocular infection or ocular inflammation in the past 2 months
* Any abnormality preventing reliable fluorophotometry of either eye,such as corneal scarring or severe dry eye that results in punctuate fluorescein staining of the cornea
* Intraocular surgery within 6 months
* Serious hypersensitivity to any components of the study medications or risk from treatment with glaucoma medications, such as severe asthma or emphysema.
* Use of any glucocorticoid by any route. Subject must be washed out of the glucocorticoid for at least 2 weeks before study entry.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with established diagnosis of retinal vascular diseases (diabetic macular edema, neovascular macular degeneration, presumed ocular histoplasmosis syndrome, high myopia) who require intravitreal injection of anti-VEGF drugs such as bevacizumab, ranibizumab or aflibercept and are likely to need three monthly doses.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Uveoscleral outflow changes | 1-2 months
  The uveoscleral outflow changes will be assess at baseline prior to any anti-VEGF treatment and after the 3rd intravitreal treatment has been done.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gulati, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Truhlsen Eye Institute, Omaha, Nebraska
  - University of Nebraska Medical Center, Department of Ophthalmology and Visual Sciences, Omaha, Nebraska